CLINICAL TRIAL: NCT06457906
Title: SRS/SRT/Hypo-RT Versus HA-WBRT for No More Than 10 Brain Metastases in Patients With Small-Cell Lung Cancer: A Prospective, Randomized, Multicenter Phase III Trial (SHARP Trial)
Brief Title: SRS/SRT/Hypo-RT Versus HA-WBRT for No More Than 10 Brain Metastases in SCLC
Acronym: SHARP
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Bi Nan, Professor and Director of Thoracic Division, Department of Radiation Oncology, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCC3982
Record Dates: First submitted 2024-06-10; First posted 2024-06-13 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Small-cell Lung Cancer; Brain Metastases; SRS; Stereotactic Radiotherapy; Whole Brain Radiotherpay; Hippocampal-avoidance
Keywords: Small-cell Lung Cancer; Brain Metastases; SRS; Stereotactic radiotherapy; Whole brain radiotherpay; Hypofractionaed radiotherapy; Hippocampal-avoidance
MeSH Terms: conditions — Small Cell Lung Carcinoma; Brain Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SRS/SRT/Hypo-RT group (Experimental): The patients in this group will receive local treatment for BM.
  Interventions: Combination Product: Experimental group (SRS/SRT/Hypo-RT)
- HA-WBRT group (Active Comparator): The patients in this group will receive HA-WBRT.
  Interventions: Radiation: Controled group (HA-WBRT)

INTERVENTIONS:
Combination Product: Experimental group (SRS/SRT/Hypo-RT) — The prescription dose of SRS/SRT is 18-22Gy in 1 fraction, 27Gy in 3 fractions and 30Gy in 5 fractions. The prescription dose of Hypo-RT is 40Gy in 8 fraction. The prescription dose could be adjusted if lesions are located in brain stem when treat with SRS/SRT/Hypo-RT.
  Arms: SRS/SRT/Hypo-RT group
Radiation: Controled group (HA-WBRT) — The prescription dose of HA-WBRT is 30Gy in 10 fraction.
  Arms: HA-WBRT group

SUMMARY:
This phase III trial compares the effect of stereotactic radiosurgery and whole brain radiation therapy that avoids the hippocampus (the memory zone of the brain) for the treatment of small cell lung cancer that has spread to the brain.

DETAILED DESCRIPTION:
Small cell lung cancer (SCLC) is the most aggressive histologic subtype of lung cancer, with a predilection for early metastases. Brain metastases (BM) are a significant threat to quality of life in patients with SCLC. Stereotactic radiosurgery (SRS)/ Stereotactic Radiotherapy (SRT) is a specialized radiation therapy that delivers a single, high dose of radiation directly to the tumor and may cause less damage to the surrounding normal tissue. Thus SRS/SRT has now emerged as the preferred treatment modality, either alone or in combination with other modalities for BM. However, given the propensity for dissemination of SCLC, SRS/SRT does not appear to be a rational approach to this pathology. Recently, in selected patients, whole brain radiotherapy (WBRT) has been omitted from the initial management for BM with the aim of reducing the potential risk of delayed neurological toxicity[1-3]. Thus, the role of upfront focal treatment by means of SRS for BM from SCLC has yet to be determined

This phase III trial compares the effect of upfront local treatment (including SRS/SRT and hypofractionated radiotherapy [Hypo-RT]) and WBRT that avoids the hippocampus (the memory zone of the brain) for the treatment of no more than 10 BM in SCLC patients. The expectation is that SRS/SRT/Hypo-RT will be one of standard upfront local treatments in SCLC patients with no more than 10 BM.

Eligible patients will be 1:1 randomized to receive ether local treatment (SRS/SRT/Hypo-RT), or hippocampal-voidance WBRT. The prescription dose of SRS/SRT is 18-22Gy in 1 fraction, 27Gy in 3 fractions and 30Gy in 5 fractions. The prescription dose of Hypo-RT is 40Gy in 8 fraction. The prescription dose of HA-WBRT is 30Gy in 10 fraction. The prescription dose could be adjusted if lesions are located in brain stem when treat with SRS/SRT/Hypo-RT.

ELIGIBILITY:
Inclusion Criteria:

Investigators should consider these factors when selecting patients for this trial. Investigators also should consider all other relevant factors (medical and non-medical), as well as the risks and benefits of the study therapy, when deciding if a patient is an appropriate candidate for this trial.

1. Adult patients (18-80 years of age) with Eastern Cooperative Oncology Group performance status 0-2 or Karnofsky performance score ≥ 70, expected life time more than 6 months;
2. Pathologically (histologically or cytologically) proven diagnosis of small cell lung cancer within 5 years of registration. If the original histologic proof of malignancy is greater than 5 years, then pathological (i.e., more recent) confirmation is required (e.g., from a systemic or brain metastasis). Patients with de novo or recurrent small cell lung cancer are permitted;
3. No more than 10 metastatic brain lesions with ≤5 cm in largest diameter and ≤150 ml in treated volume, confirmed by a high-resolution (thickness ≤2mm) , 3-dimensional T1-weighted postgadolinium magnetic resonance imaging (MRI) brain scan within 2 weeks of study initiation. All brain metastases must be outside a 5-mm margin around either hippocampus or optic pathways.
4. Not all metastatic brain lesions are recommended or suitable for surgical resection after multidisciplinary team discussion. If part of metastatic brain lesions are resected, the patient is permitted for enrollment evaluation at least two weeks after resection; 5 Patients must have the psychological ability and general health that permits completion of the study requirements, all assessment (HVLT-R, MoCA, EORTC QLQ-C30) and required follow up (at least 6 months);

6. At least one measurable BM according to the Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) criteria; 7. Women of childbearing potential and men who are sexually active should be willing and able to use medically acceptable forms of contraception during treatment on this study and for up to 180 days after completion of all treatment to prevent pregnancy or fathering a child; 8. Written informed consent (must be available before enrolment in the trial).

Exclusion Criteria:

1. Clinical or radiologic evidence of new, untreated, and/or progressive brain metastases prior to registration;
2. Previous radiotherapy of the brain;
3. Patients can not tolerate immobilization or are with MRI contraindication (i.e., cardiac pacemaker, implanted defibrillator, certain cardiac valve replacements, certain metal implants);
4. Radiographic evidence of hydrocephalus or other architectural distortion of the ventricular system, leptomeningeal metastases, increased intracranial pressure requiring immediate depression surgery.
5. Patients who have not yet recovered from acute high-grade (≥Grade 3) toxicities of prior therapies according Common Terminology Criteria for Adverse EventsVersion5.0 (CTC 5.0);
6. Presence of other serious illnesses such as acute myocardial infarction, severe arrhythmia, or psychiatric disorders within the past 6 months;
7. Known carcinoma < 5 years ago (excluding carcinoma in situ of the cervix, basal cell carcinoma, squamous cell carcinoma of the skin) requiring immediate treatment interfering with study therapy;
8. Pregnant or lactating women;
9. Participation in another clinical study or observation period of competing trials, respectively;

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2027-08-30 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Cognitive function scores | At 6 months after radiotherapy.
  Hopkins Verbal Learning Test-Revised (HVLT-R) total recall score at 6 months after radiotherapy
Meadian OS time | Measured at months 3, 6, 9, 12, 15,18, 21, 24, 30, 36,42,48,60 months after radiotherapy
  The time that half of enrolled patients died.

SECONDARY OUTCOMES:
Cognitive function scores | Measured at months 3, 6, 9, 12months after radiotherapy
  The Montreal cognitive assessment (MoCA) score at 3 ,6,9,12 months after radiotherapy
Scores of quality of life | Measured at months 3, 6, 9, 12months after radiotherapy
  The European organization for Research and Treatment of Cancer Quality of Life Questionnaire 30 (EORTC QLQ-C30) score at 3,6,9,12 months after radiotherapy
The time of neurological progression free survival | Measured at months 3, 6, 9, 12months after radiotherapy
  The time that ≥3 points reduced of HVLT-R total recall score or MoCA score after radiotherapy
The time of intracranial overall progression free survival | Measured at months 3, 6, 9, 12, 15,18, 21, 24, 30, 36,42,48,60 months after radiotherapy
  The time that half of enrolled patients had intracranial relapse
The time of overall progression free survival | Measured at months 3, 6, 9, 12, 15,18, 21, 24, 30, 36,42,48,60 months after radiotherapy
  The time that half of enrolled patients had relapse
The rate and grade of treatment related toxicity | Measured at months 3, 6, 9, 12, 15,18, 21, 24, 30, 36,42,48,60 months after radiotherapy
  All adverse events of enrolled patients after radiotherapy evaluated by CTCAE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Nan Bi, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Yomo S, Hayashi M. Upfront stereotactic radiosurgery in patients with brain metastases from small cell lung cancer: retrospective analysis of 41 patients. Radiat Oncol. 2014 Jul 8;9:152. doi: 10.1186/1748-717X-9-152. PMID 25005424
- [Background] Rusthoven CG, Yamamoto M, Bernhardt D, Smith DE, Gao D, Serizawa T, Yomo S, Aiyama H, Higuchi Y, Shuto T, Akabane A, Sato Y, Niranjan A, Faramand AM, Lunsford LD, McInerney J, Tuanquin LC, Zacharia BE, Chiang V, Singh C, Yu JB, Braunstein S, Mathieu D, Touchette CJ, Lee CC, Yang HC, Aizer AA, Cagney DN, Chan MD, Kondziolka D, Bernstein K, Silverman JS, Grills IS, Siddiqui ZA, Yuan JC, Sheehan JP, Cordeiro D, Nosaki K, Seto T, Deibert CP, Verma V, Day S, Halasz LM, Warnick RE, Trifiletti DM, Palmer JD, Attia A, Li B, Cifarelli CP, Brown PD, Vargo JA, Combs SE, Kessel KA, Rieken S, Patel S, Guckenberger M, Andratschke N, Kavanagh BD, Robin TP. Evaluation of First-line Radiosurgery vs Whole-Brain Radiotherapy for Small Cell Lung Cancer Brain Metastases: The FIRE-SCLC Cohort Study. JAMA Oncol. 2020 Jul 1;6(7):1028-1037. doi: 10.1001/jamaoncol.2020.1271. PMID 32496550
- [Background] Robin TP, Jones BL, Amini A, Koshy M, Gaspar LE, Liu AK, Nath SK, Kavanagh BD, Camidge DR, Rusthoven CG. Radiosurgery alone is associated with favorable outcomes for brain metastases from small-cell lung cancer. Lung Cancer. 2018 Jun;120:88-90. doi: 10.1016/j.lungcan.2018.03.027. Epub 2018 Apr 2. PMID 29748022